CLINICAL TRIAL: NCT05312177
Title: Congenital Heart Disease: Impact on Learning and Development in Down Syndrome (CHILD-DS)
Acronym: CHILD-DS
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: CHILD-DS; 3U24HL135691-03S1 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2022-04-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-10

CONDITIONS: Down Syndrome; Congenital Heart Disease
Keywords: Down Syndrome; CHD; Congenital Heart Disease; Pediatric Heart Network; INCLUDE
MeSH Terms: conditions — Down Syndrome; Heart Defects, Congenital | interventions — Reoperation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We aim to collect saliva samples from study participants during the single study visit at the PHN site, which will be preserved and processed by the PHN Biorepository for DNA storage for future targeted research studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DS with CAVSD Repair: Children ages 5 through 12 years with Down syndrome who had Complete atrioventricular septal defect (CAVSD) repair in the first year of life and their parent(s) will be administered the Stanford-Binet Intelligence Scales, Fifth Edition (SB-5), Peabody Picture Vocabulary Test, Fifth Edition (PPVT-5), Expressive Vocabulary Test, Third Edition (EVT-3), Leiter International Performance Scale, Third Edition (Leiter-3), Vineland-3 Q-global Comprehensive Report (Vineland-3) ,Social Communication Questionnaire, Current version (SCQ), Aberrant Behavior Checklist, Second Edition, (ABC-2) and Repetitive Behavior Scale, Revised (RBS-R)
  Interventions: Other: Stanford Binet Intelligence Scales, Fifth Edition; Other: Vineland Adaptive Behavior Scales Third Edition; Other: Peabody Picture Vocabulary Test, Fifth Edition; Other: Expressive Vocabulary Test, Third Edition; Other: Leiter International Performance Scale, Third Edition; Other: Social Communication Questionnaire, Current Form; Other: Aberrant Behavior Checklist; Other: Repetitive Behavior Scale, Revised
- DS without major CHD: Children ages 5 through 12 years with Down syndrome without major Congenital Heart Disease(CHD) and their parent(s) will be administered the Stanford-Binet Intelligence Scales, Fifth Edition (SB-5), Peabody Picture Vocabulary Test, Fifth Edition (PPVT-5), Expressive Vocabulary Test, Third Edition (EVT-3), Leiter International Performance Scale, Third Edition (Leiter-3), Vineland-3 Q-global Comprehensive Report (Vineland-3) ,Social Communication Questionnaire, Current version (SCQ), Aberrant Behavior Checklist, Second Edition, (ABC-2) and Repetitive Behavior Scale, Revised (RBS-R)
  Interventions: Other: Stanford Binet Intelligence Scales, Fifth Edition; Other: Vineland Adaptive Behavior Scales Third Edition; Other: Peabody Picture Vocabulary Test, Fifth Edition; Other: Expressive Vocabulary Test, Third Edition; Other: Leiter International Performance Scale, Third Edition; Other: Social Communication Questionnaire, Current Form; Other: Aberrant Behavior Checklist; Other: Repetitive Behavior Scale, Revised

INTERVENTIONS:
Other: Stanford Binet Intelligence Scales, Fifth Edition — The SB-5 is a comprehensive measure of cognitive and intellectual functioning for individuals from age two through 85 years of age. The SB-5 individually assess a child's functioning in five areas of cognitive functioning: Fluid Reasoning, Knowledge, Quantitative Reasoning, Visual Spatial, and Working Memory. The SB-5 is well established in the existing research literature as an assessment tool to evaluate developmental and intellectual abilities in children with ND disorders.
  Other Names: SB-5
Other: Vineland Adaptive Behavior Scales Third Edition — The VABS-3 are a parent report, interview style measure of adaptive behavior for individuals ages birth through 90 months. The VABS-3 assesses adaptive behavior in four broad domains of Communication, Daily Living Skills, Socialization, and Motor Skills, and includes a Maladaptive Behavior Domain that assesses problem behaviors.
  Other Names: VABS-3
Other: Peabody Picture Vocabulary Test, Fifth Edition — The PPVT-5 is a norm-referenced language measure that evaluates single-word receptive vocabulary. The PPVT-5 provides standard scores for individuals ages 2.6 through 90 years.
  Other Names: PPVT-5
Other: Expressive Vocabulary Test, Third Edition — The EVT-3 is a norm-referenced language measure that evaluates single-word expressive vocabulary. The EVT-3 provides standard scores for individuals ages 2.6 through 90 years.
  Other Names: EVT-3
Other: Leiter International Performance Scale, Third Edition — The Leiter-3 is a nonverbal measure of cognitive functioning and fluid reasoning skills in individuals ages 3 through 75 years. The Leiter-3 measures nonverbal IQ across four subscales, including Sequential Order (SO), Form Completion (FC), Classification and Analogies (CA), and Figure Ground (FG).
  Other Names: Leiter-3
Other: Social Communication Questionnaire, Current Form — The SCQ is a parent-report measure of social communication, social interactions, play, and behavior.
  Other Names: SCQ
Other: Aberrant Behavior Checklist — The ABC-2 is a parent report measure of problematic behavior at home and in the community. It measures behavior on five subscales (1) Irritability, (2) Social Withdrawal, (3) Stereotypic Behavior, (4) Hyperactivity/Noncompliance, and (5) Inappropriate Speech.
  Other Names: ABC-2
Other: Repetitive Behavior Scale, Revised — The RBS-R is a parent report measure that comprehensively surveys for the presence of repetitive behaviors.
  Other Names: RBS-R

SUMMARY:
The study objective is to compare neurodevelopmental (ND) and behavioral outcomes between children with Down syndrome (DS) who had complete atrioventricular septal defect (CAVSD) repair and children from the same clinical sites with DS without major congenital heart disease (CHD) requiring previous or planned CHD surgery.

DETAILED DESCRIPTION:
We are conducting a multicenter cohort study, ancillary to the Pediatric Heart Network (PHN) Residual Lesion Score (RLS) study, to investigate determinants of ND and behavioral outcomes in children with DS, focusing on the role of CHD surgery. We are including children with DS who had CAVSD repair, as this group comprises 91% of all children with DS in the RLS Study, with similar underlying congenital cardiac defect and surgical repair complexity, allowing our children with DS and CHD to be a homogeneous group. Moreover, one in five individuals with DS is born with an AVSD, a 2000 times higher incidence than in those with normal chromosomes. In addition to recruiting children with DS who had CAVSD repair, we will recruit similarly-aged children with DS who do not have documented major CHD (i.e., CHD requiring previous or planned CHD surgery) to come into the same PHN site for a single study visit consisting of detailed phenotyping by completion of a Health & Developmental History Intake form, ND and behavioral assessments, and optional collection and storage of saliva specimens in the PHN Biorepository. By building our sample from RLS Study participants and recruiting additional children who had infant CAVSD repair and meet study eligibility criteria, as well as a comparison group from the same PHN sites, we are leveraging rich prospective data in a group of DS children with CAVSD repair from a nationally representative sample, and the expertise of the PHN and Boston Children's Hospital (BCH).

ELIGIBILITY:
Inclusion Criteria:

Down Syndrome CAVSD Repair Group:

* Trisomy 21
* Male or Female, ages 5 years through 12 years
* Had CAVSD repair within the first year of life
* Parent or guardian and patient willing to comply with protocol and complete all study assessments; parent or guardian willing to provide written informed consent
* Child able to speak and understand English

Down Syndrome Comparison Group

* Trisomy 21
* Male or Female, age 5 years through 12 years
* No major CHD, defined as CHD requiring previous or planned CHD surgery
* Parent or guardian and patient willing to comply with protocol and complete all study assessments; parent or guardian willing to provide written informed consent
* Child able to speak and understand English

Exclusion Criteria:

Both Groups

- Mosaic DS

Down Syndrome CAVSD Repair Group only - Did not have CAVSD repair in the first year of life

Down Syndrome Comparison Group only

- Major CHD requiring previous or planned CHD surgery - i.e., CHD surgery occurring (a) in the period between birth and time of recruitment into the CHILD-DS Study, or (b) planned for a future date.

Ages: 60 Months to 155 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: PHN RLS Study participants with DS and CAVSD repair from the PHN sites are eligible to participate in this study. Children with a diagnosis of mosaic DS will be excluded, as these forms of DS show different ND trajectories and are usually excluded. While data on mosaic DS were not collected in the RLS Study, we anticipate few if any to have this diagnosis. The DS comparison group will be required to have no major CHD, defined as CHD that requires CHD surgery (a) in the period between birth and recruitment into the CHILD-DS Study or (b) planned for a future date.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcomes between children with DS who had CAVSD repair and children from the same clinical sites with DS without major CHD. | 1 day
  Verbal and non-verbal ratio intelligent quotients (IQs) derived from the Stanford Binet Intelligence Scales will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.
Behavioral outcomes between children with DS who had CAVSD repair and children from the same clinical sites with DS without major CHD. | 1 day
  Adaptive composite scores from the Vineland Adaptive Behavior Scales will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.
Language abilities compared between the children with DS and CAVSD repair and the children with DS without major CHD. | 1 day
  Using the Peabody Picture Vocabulary Test, Expressive Vocabulary Test, and Leiter International Performance Scale total language, auditory comprehension, and expressive communication will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.
Emotional outcomes compared between the children with DS and CAVSD repair and the children with DS without major CHD. | 1 day
  Using the Repetitive Behavior Scale and Aberrant Behavior Checklist , behavioral and emotional problems will be compared will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.
Social Communication compared between the children with DS and CAVSD repair and the children with DS without major CHD. | 1 day
  Using the Social Communication Questionnaire, social communication, social interactions, play and behavior will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.

SECONDARY OUTCOMES:
Comorbidities as predictors of neurodevelopment and behavior | 1 day
  Comorbidities will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.
Sociodemographic factors as predictors of neurodevelopment and behavior | 1 day
  Sociodemographic factors, such as will be compared between the children with DS and CAVSD repair and the children with DS without major CHD.

CONTACTS AND LOCATIONS:
Overall Officials: Maria VanRompay, PhD, Principal Investigator — Carelon Research
Locations (14):
- United States (13):
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System/Mott Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia College of Physicians and Surgeons, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Public Use Datasets are created after study closeout and are made available on the PHN public website. Annotated study data collection forms, Statistical Analysis Program (SAS) datasets, and excel datasets are made available, as well as de-identified study cohort characteristics.
Supporting Information: Study Protocol, ICF
Time Frame: Data is available one year after study closeout and is available indefinitely.
Access Criteria: log-in and password
URL: https://www.pediatricheartnetwork.org/login/